CLINICAL TRIAL: NCT01545596
Title: A Randomized Effectiveness Trial of Early Hemodynamic Support in Patients Demonstrating a Double and Triple Low Combination of Mean Arterial Pressure, and Either End-tidal Anesthetic Concentration or Bispectral Index.
Brief Title: Will a Real Time Advisory for Double Low State Change Clinical Behavior and Impact Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GCO 10-0111; HSM 11-00590
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Ability to Influence Behavior; Information Systems
Keywords: Intraoperative Monitoring; Decision Support Systems; anesthesia outcomes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Notification Group (Experimental): Anesthesia team receives notification when a double low condition exists. The anesthesia team makes a decision to intervene or not.
  Interventions: Behavioral: Notification Group
- No Notification (No Intervention): No additional notification given to anesthesia team apart from the information on their monitors.

INTERVENTIONS:
Behavioral: Notification Group — Anesthesia team receives notification when a double low condition exists. The anesthesia team makes a decision to intervene or not.
  Other Names: Notification through anesthesia system
  Arms: Notification Group

SUMMARY:
The objective of this study is to use a decision-support system combined with an electronic anesthesia record to detect double low clinical conditions (Mean Arterial Pressure (MAP) < 75 mmHg, and Bispectral Index (BIS) < 45) and generate alerts suggesting hemodynamic support. Specifically, the project will test the hypothesis that providing Double Low alerts reduces 90-day mortality. Secondary outcomes will be the fraction of alerts that generate early clinician responses, subsequent changes in MAP and hospital length of stay.

DETAILED DESCRIPTION:
Data that is routinely collected as part of standard of care intraoperative monitoring including blood pressure, amount of anesthetic administered and a form of processes electroencephalogram called the bispectral index, which is a measure of depth of anesthesia all enter in an electronic record keeper. This project monitors for a combination of a blood pressure below mean of 75mmHg and a BIS of 45. When this is detected, half of the anesthesiologists caring for patients receive a text message on the computer screen and their pagers indicating that a double low situation exists and that they should consider intervening. The other half of practitioners are not provided with the additional messages, although all of the same information is available in the operating room (OR). Most patients undergoing general non-cardiac anesthesia at Mount Sinai are eligible. Documentation of consent was waived. All patients are informed of the ongoing project upon admission and are given a variety of methods of opting out of the project.

The analysis seeks to determine if the messages were effective at influencing clinician behavior and whether that change would make a difference in either length of stay or 90 day mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for general anesthesia and have BIS monitors

Exclusion Criteria:

* patients who opt out of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20237 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mortality | at 90 days

SECONDARY OUTCOMES:
Response to Notification | Intraoperative
  proportion of anesthesia teams that respond to a double low event with either a vasopressor or decrease in the dose of volatile anesthetic
Effect of response | Intraoperative
  An evaluation as to whether the response elicited resulted in less double low physiology

CONTACTS AND LOCATIONS:
Overall Officials: David Reich, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] McCormick PJ, Levin MA, Lin HM, Sessler DI, Reich DL. Effectiveness of an Electronic Alert for Hypotension and Low Bispectral Index on 90-day Postoperative Mortality: A Prospective, Randomized Trial. Anesthesiology. 2016 Dec;125(6):1113-1120. doi: 10.1097/ALN.0000000000001296. PMID 27775995